CLINICAL TRIAL: NCT06942637
Title: Effectiveness of Integrated Network for Student Psychosocial Intervention, Resilience, and Education (INSPIRE) on Mental Health Outcomes Among Indonesian Adolescents in Bandung: A Randomised Controlled Trial and Process Evaluation
Brief Title: Effectiveness of Integrated Network for Student Psychosocial Intervention, Resilience, and Education (INSPIRE) on Mental Health Outcomes Among Indonesian Adolescents in Bandung
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Indonesia Endowment Fund for Education (LPDP), Republic of Indonesia (Unknown)
Responsible Party: Principal Investigator, Shefaly Shorey, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 241/UN6.KEP/EC/2025
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Adolescents; Health Knowledge; Mental Health; Health Literacy; Resilience; Depression; Anxiety; Parents; School Intervention
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Two-group parallel-armed randomized controlled trial (RCT) with a pretest and repeated posttest experimental design. Sample size was determined via power analyses informed by three adolescent mental health intervention studies (Casañas et al., 2022; Kaligis et al., 2023; Liddle et al., 2021). Reported effects ranged from small-to-medium (d = 0.26; Liddle) to medium-to-large (d = 0.64; Kaligis), with Casañas reporting 0.382-0.705. To ensure conservative estimates, calculations used the smallest effect (d = 0.26). A two-tailed test (α = 0.05, power = 0.80) indicated 230 participants per arm. Adjusting for 32% attrition, the final target sample size was set at 340 per arm (N = 680).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard school health routine care (No Intervention)
- INSPIRE Intervention (Experimental): Receive an 8-week school-based program aimed at enhancing adolescent mental health, attitudes towards mental health and help-seeking behaviors, mental health literacy, resilience and addressing depression and anxiety.
  Interventions: Behavioral: INSPIRE (Integrated Network for Student Psychosocial Intervention, Resilience, and Education)

INTERVENTIONS:
Behavioral: INSPIRE (Integrated Network for Student Psychosocial Intervention, Resilience, and Education) — The INSPIRE intervention is an 8-week school-based program aimed at enhancing adolescent mental health, attitudes towards mental health and help-seeking behaviors, mental health literacy, resilience and addressing depression and anxiety. Trained school counsellors deliver this structured curriculum using comprehensive materials including lesson plans, activities, and visual aids. the program provides supplementary resources for both participating students and their parents .
  Arms: INSPIRE Intervention

SUMMARY:
The INSPIRE (Integrated Network for Student Psychosocial Intervention, Resilience, and Education) intervention is an 8-week, school-based mental health program designed to enhance adolescents' mental health literacy and resilience while addressing symptoms of depression and anxiety. Implementation is conducted by school counselors who undergo an intensive two-day training program. The intervention is supported by comprehensive curriculum materials including detailed lesson plans, activities, discussion prompts, and instructional slides featuring key concepts, visuals, and explanatory content. Supplementary materials are developed for both participating adolescents and their parents.

The study aims to:

1. Evaluate the usability and feasibility of the INSPIRE intervention within the school environment.
2. Assess the intervention's effectiveness in improving:

   * Primary outcome: Mental health knowledge among adolescents
   * Secondary outcomes: Attitudes toward mental health, help-seeking behaviors, mental health literacy, resilience, and symptoms of depression and anxiety among adolescents
   * Secondary outcomes: mental health knowledge, attitudes, help-seeking behaviors, and mental health literacy among parents
3. Explore the experiences of intervention participants (both adolescents and parents) against the control group to develop comprehensive insights into the psychosocial intervention's impact.

The research hypothesis proposes that the INSPIRE intervention group will demonstrate significantly higher scores in mental health knowledge, more positive attitudes toward mental health, increased help-seeking behaviors, enhanced mental health literacy, and greater resilience, while simultaneously showing reduced symptoms of depression and anxiety compared to the control group receiving standard care. These outcomes will be measured immediately following the intervention (post-test 1) and at one-month follow-up (post-test 2).

DETAILED DESCRIPTION:
Pilot Study The pilot study was conducted as a two-centre, two-arm cluster randomised controlled trial with a pre-test-post-test design and a 1:1 allocation ratio. Randomisation was performed at the school (cluster) level to minimise contamination. The pilot phase was implemented from 28 April to July 2025.

Randomised Controlled Trial (RCT) The full-scale randomised controlled trial expanded to a multi-centre design involving five centres, maintaining a two-arm cluster randomised structure with school-level allocation. The RCT commenced in September 2025 and is currently ongoing.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for adolescents are as follows:

* Unmarried, 13-15 years old, school-going, healthy adolescents enrolled in an Indonesian public junior high school
* Able to read, understand, and converse in Bahasa Indonesia.

The inclusion criteria for parents are as follows:

* The biological father, mother, or an adult who fulfils a parental or guardian role for the participating adolescent
* Able to understand and communicate in Bahasa Indonesia.

Exclusion Criteria:

* Adolescents who are working, clinically diagnosed with severe mental disorders, such as schizophrenia or psychosis, at high risk for mental health disorders (e.g., teenage pregnancy), or are cognitively impaired will be excluded.
* Parents with severe mental disorders or cognitive impairment that may hinder participation will be excluded.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 680 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Adolescents' mental health knowledge | Immediately following the intervention (post-test 1)
  13-item mental health knowledge scale. Total scores range from 0 to 13, with higher scores indicating better mental health knowledge.
Adolescents' mental health knowledge | At one-month follow-up (post-test 2).
  13-item mental health knowledge scale. Total scores range from 0 to 13, with higher scores indicating better mental health knowledge.

SECONDARY OUTCOMES:
Adolescents' attitudes towards mental health | immediately following the intervention (post-test 1)
  12-item attitude toward mental health scale. Scores range from 12 to 60, with higher scores indicating more positive attitudes.
Adolescents' attitudes towards mental health | At one-month follow-up (post-test 2).
  12-item attitude toward mental health scale. Scores range from 12 to 60, with higher scores indicating more positive attitudes.
Adolescents' attitudes toward help-seeking behaviors | Immediately following the intervention (post-test 1)
  5-item attitude toward mental help-seeking behaviors questionnaire. Scores range from 5 to 15, with higher scores indicating more positive attitudes toward help-seeking behaviors.
Adolescents' attitudes toward help-seeking behaviors | At one-month follow-up (post-test 2).
  5-item attitude toward mental help-seeking behaviors questionnaire. Scores range from 5 to 15, with higher scores indicating more positive attitudes toward help-seeking behaviors.
Adolescents' mental health literacy | Immediately following the intervention (post-test 1)
  the 50-item Knowledge and Attitudes to Mental Health Scales, with total scores ranging from 0 to 200. Higher scores indicated higher mental health literacy.
Adolescents' mental health literacy | At one-month follow-up (post-test 2).
  the 50-item Knowledge and Attitudes to Mental Health Scales, with total scores ranging from 0 to 200. Higher scores indicated higher mental health literacy.
Adolescents' resilience | Immediately following the intervention (post-test 1)
  the nine-item resilience evaluation scale, with the total scores ranging from 0 to 36. Higher scores indicated higher psychological resilience.
Adolescents' resilience | At one-month follow-up (post-test 2).
  the nine-item resilience evaluation scale, with the total scores ranging from 0 to 36. Higher scores indicated higher psychological resilience.
Adolescents' depression | Immediately following the intervention (post-test 1)
  the nine-item Patient Health Questionnaire, with total scores ranging from 0 to 27. Higher scores indicate more severe depressive symptoms.
Adolescents' depression | At one-month follow-up (post-test 2).
  the nine-item Patient Health Questionnaire, with total scores ranging from 0 to 27. Higher scores indicate more severe depressive symptoms.
Adolescents' anxiety | Immediately following the intervention (post-test 1)
  the 7-item Generalized Anxiety Disorder scale, with total scores ranging from 0 to 21. Higher scores indicate more severe anxiety symptoms.
Adolescents' anxiety | At one-month follow-up (post-test 2).
  the 7-item Generalized Anxiety Disorder scale, with total scores ranging from 0 to 21. Higher scores indicate more severe anxiety symptoms.
Parents' mental health knowledge | Immediately following the intervention (post-test 1)
  13-item mental health knowledge scale. Total scores range from 0 to 13, with higher scores indicating better mental health knowledge.
Parents' mental health knowledge | At one-month follow-up (post-test 2).
  13-item mental health knowledge scale. Total scores range from 0 to 13, with higher scores indicating better mental health knowledge.
Parents' attitudes towards mental health | immediately following the intervention (post-test 1)
  12-item attitude toward mental health scale. Scores range from 12 to 60, with higher scores indicating more positive attitudes.
Parents' attitudes towards mental health | At one-month follow-up (post-test 2).
  12-item attitude toward mental health scale. Scores range from 12 to 60, with higher scores indicating more positive attitudes.
Parents' attitudes toward help-seeking behaviors | Immediately following the intervention (post-test 1)
  5-item attitude toward mental help-seeking behaviors questionnaire. Scores range from 5 to 15, with higher scores indicating more positive attitudes toward help-seeking behaviors.
Parents' attitudes toward help-seeking behaviors | At one-month follow-up (post-test 2).
  5-item attitude toward mental help-seeking behaviors questionnaire. Scores range from 5 to 15, with higher scores indicating more positive attitudes toward help-seeking behaviors.
Parents' mental health literacy | Immediately following the intervention (post-test 1)
  The 16-item Mental Health Literacy Questionnaire, with total scores ranging from 16 to 80. Higher scores indicated higher mental health literacy.
Parents' mental health literacy | At one-month follow-up (post-test 2).
  The 16-item Mental Health Literacy Questionnaire, with total scores ranging from 16 to 80. Higher scores indicated higher mental health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandung City Education Office and Junior high schools (Sekolah Menengah Pertama), Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No